CLINICAL TRIAL: NCT02769182
Title: Development and Validation of a Smart Phone Based System to Enhance Gait, Cognition and Socialization in Elderly Fallers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: HIT Holon Institute of Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-13-NG-127-CTIL
Record Dates: First submitted 2016-05-02; First posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Older Adults
Keywords: Older adults; falls; cognition; smart phone
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring and training using the system (Experimental)
  Interventions: Device: Monitoring and training using the system
- Standard of care (Active Comparator)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Device: Monitoring and training using the system — subjects and caregivers will be trained on using the system and receive a 'user manual' delineating all procedures and possible applications of the system, as well as operations for daily charging of the sensors and smart phone. They will then be fitted with the sensors. The clinician will set all necessary applications, including setting the cognitive games application and the 'network of users'. Users and care givers will be informed of the personalized recommendations system that will provide the user with daily feedback on activity and weekly recommendations and goals for duration of the study. A helpline will be provided in case technological problems occur or for routine support.
  Arms: Monitoring and training using the system
Behavioral: Standard of care — Subjects in this group will not receive the system but will encouraged to continue with their daily living routine and provided with recommendations for stretching and strengthening exercises. The control group subjects will be assessed at the same three time points as those in the experimental group. Subjects in both groups will also receive written information about the importance of activity, cognitive enhancing tasks, avoidance of falls and home hazards. In Israel, this information combined with an exercise prescription is considered the 'standard of care' for community-dwelling older adults.
  Arms: Standard of care

SUMMARY:
The main objective of this research is to develop and validate a technology-based solution that addresses the diminished mobility, increased fall risk and impaired cognitive function that are so common among older adults, enabling them to live longer successfully and independently.

DETAILED DESCRIPTION:
A comprehensive system will be developed to promote mobility, enhance cognitive function, reduce sedentary behavior, increase independence and encourage social inclusion. This novel system will have two distinct yet complementary features: monitoring and treatment that will serve as an "all in one system". The system will consist of wearable sensors and a proprietary developed application. The wearable inertial sensors will measure the acceleration and orientation of the feet during movement. The sensors will feed real-time data to the system, which will process this data using a set of proprietary algorithms enabling continuous monitoring of activity, gait and fall risk, and independence. In addition, designated applications for direct cognitive assessment and training of older adults in their home and community environment will also be used via the Smart phone or mobile tablet. The training, both physical and cognitive, will also include multi-user interactions .Data collected by the system will be processed and integrated to provide comprehensive feedback from multiple domains to the user, caregiver and clinician by way of recommendations and personalized treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 65-85 years
* History of 1 fall or more in the year prior to the study.

Exclusion Criteria:

* Signs of dementia : Montreal Cognitive Assessment (MoCa) <21 and/or mini mental state examination(MMSE) <24.
* Psychiatric co-morbidities :major depression as determined by Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria
* Co-existing somatic disorders
* History of stroke
* Neurologic disorders that interferes with normal walking (e.g., Parkinson's disease or Alzheimer's disease),
* Cannot walk without assistance,
* Severe head trauma or brain tumor,
* Severe hearing or visual loss (determined by the visual acuity test),
* Cardio-vascular contradictions (as determined by a physician),
* Inability to use a Smart phone because of visual and manual impairment or have unstable medical conditions.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in average number of steps per day | Number of steps will be measured during one week after each assessment - at baseline, immediately after the training and 3 months after the training.
  This will be evaluated by a small, lightweight waterproof accelerometer placed on the lower back of the participants (Axivity Ltd.)
Changes in the color Trails Making Test part B | At baseline, immediately after the training and 3 months after completing the training.

SECONDARY OUTCOMES:
Changes in gait speed | At baseline, immediately after the training and 3 months after completing the training.
  gait speed will be evaluated under two conditions each over 1 minute: i) walking at comfortable speed, ii) walking while performing a cognitive task (dual task).
Changes in fear of falling | At baseline, immediately after the training and 3 months after completing the training
  falls Efficacy Scale International (FES-I).
Changes in endurance | At baseline, immediately after the training and 3 months after completing the training
  Total distance walked in six minutes (6MWT).
Changes in social connectedness | At baseline, immediately after the training and 3 months after completing the training
  Social engagement: the Berkman-Syme Social Network Index
Changes in cognitive function: score in Frontal Assessment Battery | At baseline, immediately after the training and 3 months after completing the training
  Frontal Assessment Battery: this battery is sensitive to frontal lobe dysfunction consists of six subtests exploring the following: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. It takes approximately 10 minutes to administer.
Changes in functional mobility: dynamic gait index (DGI) score | At baseline, immediately after the training and 3 months after completing the training
  DGI is a clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks
Changes in the Short Form Health Survey | At baseline, immediately after the training and 3 months after completing the training
  The Short Form Health Survey to evaluate different dimensions of health related quality of life including mobility, emotional well-being, and cognitive impairment.
Changes in stride length | At baseline, immediately after the training and 3 months after completing the training.
  Stride length will be evaluated under two conditions each over 1 minute: i) walking at
Changes in stride and swing time variability | At baseline, immediately after the training and 3 months after completing the training.
  Stride and swing time variability will be evaluated under two conditions each over 1 minute: i) walking at
Changes in cognitive function: number of digits | At baseline, immediately after the training and 3 months after completing the training
  Working memory (forward and backward digit span): Forward and backward digit span is a common measure of short-term memory (working memory). It is also a component of cognitive ability tests. Backward memory span is a more challenging variation which involves recalling items in reverse order.
Changes in cognitive function: number of correct / incorrect answers | At baseline, immediately after the training and 3 months after completing the training
  Dual tasking (DT) walking performance: alternation in the ability to walk while simultaneously performing another task, have been related to gait and balance impairment. The negative effects of DT have been associated with an increased risk of falling, underscoring the clinical importance of DT abilities
Changes in functional mobility: score in Four Square Step Test | At baseline, immediately after the training and 3 months after completing the training
  Four Square Step Test is a dynamic balance test that clinically assesses the person's ability to step over objects forward, sideways, and backwards

IPD SHARING:
Plan to Share IPD: No